CLINICAL TRIAL: NCT04089306
Title: Integration of Palliative Care in an Oncology and Hematology Unit : a Retrospective Monocentric Study
Brief Title: Integration of Palliative Care in an Oncology and Hematology Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7424
Record Dates: First submitted 2019-04-23; First posted 2019-09-13 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-04

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; End of Life; Agressiveness of Care; Palliative Care integration
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main goal of this study is to assess retrospectively the integration of Palliative Care in an oncology and hematology unit. The investigators will study the last six month of life on advanced cancer patients and retrieve data from their medical file to obtain criterias of quality of care and integration of palliative care in this population.

Those criterias have been used before in other setting (Earle Criterias, ESMO Recommendations) and The investigators will compare our data to existing publications.

They also hope to see if it is retrospectively possible to assess the probability of death using the Pronopall score. This will help them asses if aggressive end of life care could have been avoided using the Pronopall Score

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Patient who has been followed in the oncohematology Unit of the University Hospital of Strasbourg for a solid tumor or haematological cancer
* Died within the 1rst of January 2017 and the 31st of December 2018
* The patient has not expressed an opposition to the use of his medical data during his lifetime.

Exclusion Criteria:

* Patient receiving allogeneic stem cell transplant
* Patient expressed during his lifetime an opposition regarding the use of his medical data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who has been followed in the oncohematology Unit of the University Hospital of Strasbourg for a solid tumor or haematological cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of palliative care in oncohematology department | The period from January 1st, 2017 to December 31, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Hematologie Et D'Oncologie, Strasbourg, France